CLINICAL TRIAL: NCT04529369
Title: Efficacy and Long-term Durability of Middle Lobe Only (MLO) Versus Complete Trans-Urethral Vaporization of the Prostate (PVP), Prospective Cohort Study.
Brief Title: Middle Lobe Only Laser Vaporization or Total Prostate Vaporization of the Prostate, Prospective Cohort Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Jacques Corcos, Professor of Surgery (Urology), Jewish General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MP-05-2021-2448 (MP)
Record Dates: First submitted 2020-08-18; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prominent middle lobe BPH satisfactory channel after MLO PVP (Experimental)
  Interventions: Procedure: Middle lobe only Photoselective vaporization of the prostate (PVP)
- Prominent middle lobe BPH unsatisfactory channel after MLO PVP (Active Comparator)
  Interventions: Procedure: Complete PVP

INTERVENTIONS:
Procedure: Middle lobe only Photoselective vaporization of the prostate (PVP) — Middle lobe only Photoselective vaporization of the prostate (PVP) without vaporization of the lateral lobes
  Arms: Prominent middle lobe BPH satisfactory channel after MLO PVP
Procedure: Complete PVP — Traditional Photoselective vaporization of the prostate PVP
  Arms: Prominent middle lobe BPH unsatisfactory channel after MLO PVP

SUMMARY:
The investigator aims to prospectively investigate the efficacy and durability of the middle lobe only versus traditional complete photoselective greenlight vaporization of the prostate in patients with prominent middle lobe. The investigator will select patients based on pre-op cystoscopy if patients have a prominent middle lobe to participate in this study. Researches will start to vaporize only the middle lobe then, at the end of this step, The investigator will look at the verumontanum into the prostatic fossa and determine if the patient is having adequate opened prostatic fossa or not. Patients with unsatisfactory opened fossa will have a complete PVP of lateral lobes, while patients with a satisfactory channel will not receive a complete PVP. Primary objectives of the study are to look into pre and post-operative uroflowmetry and post-void residual, International prostate symptoms scores, need of catheterization, and need for secondary interventions over five then ten years. Secondary objectives are to look into erectile and ejaculatory status using the Male Sexual Health Questionnaire (MSHQ) and MSHQ-EjD Short Form for Assessing EjD. Researchers will follow the patients at three months, six months, one year then yearly for five years then an extension to up to 10 years.

DETAILED DESCRIPTION:
Introduction:

Transurethral resection of the prostate (TURP) is considered the treatment of choice for patients suffering from benign prostatic hyperplasia (BPH) refractory to medical treatments or in patients with refractory urinary retention (1). It involves complete resection of the transitional zone of the prostate from the verumontanum to the bladder neck (2). Classical TURP has a high risk of ejaculatory dysfunction (65-70%) (2), and a 7% to 13% risk of bleeding that requires transfusion (3). To reduce these complications, newer technologies have been introduced to lower these associated risks, such as greenlight laser, Rezum, and Urolift (1).

The dynamic of bladder outlet obstruction related to BPH adenoma site and distribution has not been completely elucidated. In a study that looked into this relationship, it suggested that the presence of intravesical prostatic protrusion (IPP) has been associated with the presence of prostatic adenoma with high sensitivity (95.4%), a high specificity (100%), and a high positive predictive value (100%), with the negative predictive value of (50%). Furthermore, the mean maximum flow rate (Qmax) in patients with only lateral lobe prostatic adenoma evaluated by cystoscopy was 16ml/s, while patients with middle lobe only adenoma have a flow max of 11.6 ml/s. When patients have both middle and lateral lobes, the mean Qmax was 8.9 ml/sec (4). These findings highlight the major role of middle lobe adenoma and intravesical prostatic protrusion (which is usually an extension of the middle lobe), into the urodynamics of bladder outlet obstruction. Also, the intravesical prostatic extension has been suggested to cause a "ball-valve" effect that contributes significantly to the urodynamic bladder outlet obstruction (5). In a retrospective study, middle lobe only TURP for patients with prominent middle lobe adenoma and IPP of more than 10 mm, in patients with bothersome BPH symptoms or urinary retention, was associated with improvement in Qmax, Post-void residual and reduction of the international prostate symptoms score (IPSS), over a follow-up period up to 12 years. The urodynamic outcomes were comparable to traditional TURP results but with no change in ejaculatory bother scores pre and postoperatively. It also enabled including patients with larger prostate sizes (up to 178 g) that would require open prostatectomy or complete laser enucleation of the prostate (5).

Rationale:

Middle-lobe only TURP procedure has demonstrated durable, successful urodynamic outcomes in patients with significant bladder outlet obstruction caused by middle lobe with IPP of more than 10 mm, with no change in ejaculatory status after such procedure in retrospective fashion (5). No prospective studies have been done to document this effect. Also, the use of this procedure in patients with predominant meddle-lobe prostatic adenoma with minimal or no IPP has not been evaluated. Furthermore, the use of greenlight vaporization, which is proven to cause a significant reduction in blood loss, blood transfusion, and reduced hospital stay when compared to traditional TURP (6).

This project will investigate the efficacy and durability of laser vaporization of the middle lobe only laser vaporization of prostate in patients with middle-lobe predominant prostatic adenoma occlusion, causing bothersome lower urinary tract symptoms (LUTS) or urinary retention that are refractory to medical treatment. The results of those patients will be compared to patients who will go complete PVP.

Study Objectives:

Primary objectives:

* To determine the difference in the incidence of inability to void that needs surgical intervention after a middle lobe only PVP compared to complete PVP.
* To determine the improvement in IPSS, Qmax, and post-void residual (PVR) in patients with bladder outlet obstruction caused by middle-lobe predominant prostatic adenoma leading to refractory bothersome LUTS or urinary retention, who will undergo middle lobe only greenlight photoselective vaporization of the prostate (PVP) or complete PVP in a prospective fashion.
* Compare the difference IPSS improvement in patients who underwent Middle lobe only PVP and patients who underwent complete PVP
* To evaluate the change in ejaculatory status before and after the procedure Male Sexual Health Questionnaire to Assess Ejaculatory Dysfunction (MSHQ-EjD) and compare the scores between the groups.

Secondary Objectives:

* Subset analysis of the efficacy and change of treatment urodynamic outcomes based on prostate size, PSA, and the presence or absence of IPP and/or lateral lobe adenomas.
* Documenting of the need for additional treatment of interventions
* The documentation of the blood loss and the need for blood transfusion
* Determination of the rate of patients that initially thought to have middle lobe predominant obstruction on pre-operative cystoscopy but needed complete PVP due to inadequate removal of adenoma after completing middle-lobe only PVP
* Documentation of changes in erectile function using the Male Sexual Health Questionnaire (MSHQ)
* Determination of the need to be on BPH medication in both groups at each follow up visit.
* Documentation of the presence of dysuria and compare it between the groups.

Investigational Plan:

Overall Study Design and Plan: Description:

* We will conduct a prospective cohort study collecting patients with middle-lobe predominant prostatic adenoma causing BOO who failed medical treatment and need surgical intervention.
* Patients who tried medical treatment and have significant LUTS or urinary retention and require surgical intervention will require cystoscopy examination, PSA and ultrasound sizing of prostate as standard of care for this subset of patients.
* If the patient fits the inclusion and exclusion criteria for this study, the patient will be recruited, and he will sign an informed consent form if he agrees to participate in this study.
* We will also collect:

  1. Patient's demographic data, such as age, co-morbidities and BMI
  2. IPSS, MSHQ-EjD, and MSHQ scores.
  3. Pre-operative Q-max and PVR results.
  4. Pre-operative BPH and/or erectile dysfunction medical treatment, used prior to the surgical intervention.
  5. Pre-operative PSA, transabdominal ultrasound sizing of the prostate, serum creatinine and hemoglobin, urinalysis and culture, cystoscopy findings including the anatomical distribution of prostatic adenomas

Procedure :

* Patient will undergo Middle-Lobe only PVP procedure. At the end of the vaporization of the middle lobe, the surgeon will evaluate prostatic urethra at its distal end to evaluate the opening created into the prostate.

  1. If the endoscopic view shows absence of obstructing prostatic adenoma, the procedure will be terminated and the patient will be included in the Middle lobe only group
  2. If the endoscopic view shows significant obstruction caused by lateral prostatic lobe, completion of lateral lobes vaporization will be carried out and the patient will be included in the complete PVP group
* The postoperative stay and perioperative complications will be documented, including the postoperative hemoglobin, and the need for transfusion.
* Medical treatment discontinuation: Alpha-blockers and 5-alpha reductase inhibitors will be stopped prior to discharge for all patients.
* Investigators will document the success of the tria-of-void (TOV) prior to discharge

  1. Patients with successful TOV, the first follow up will be in 2 months as a standard of care.
  2. Patients who will have a failed TOV prior to discharge will undergo the standard of care protocol for failed TOV used in standard PVP and TURP.

  2a. Patients will be discharged home with a Foley catheter 2b. We will book a second trial of void in the clinic within 5 to 7 days after surgery 2b1. If 2nd TOV is successful, patient will be followed 2 months after the procedure as the rest of patients 2b2. If the 2nd TOV failed, we will reinsert a foley catheter and we will arrange cystoscopy to reevaluate the prostatic urethra and the bladder followed by a 3rd TOV.

  2b2a. If successful TOV, patient will be back to the regular follow up. 2b2b. If there is a significant obstruction and failed TOV, a completion PVP will suggested as a standard of care.

  2b2c. If there is no blockage and a failed TOV, patient will be given the standard options of clean intermittent catheterization, indwelling suprapubic catheter, and indwelling urethral catheter.

  2b3. The data of patients who will fail TOV and their final outcomes will be collected and reported in the study.
* Post-operative follow-up protocol for included patients will be done at 2 months post-operatively, then at 6 months, then at 1 year then yearly, after. This is like standard of care in patients after PVP. A postoperative visit will document the following:

  1. IPSS, OABSS, MSHQ-EjD and MSHQ scores in each visit
  2. Symptoms improvement and overall satisfaction with the procedure in each visit as standard of care
  3. Recurrence of any LUTS as the standard of care
  4. Presence of urine culture-proven UTI The use of any BPH or OAB medications as the standard of care
  5. The presence or resolution of dysuria as standard of care
  6. Presence or absence of Incontinence, and type of incontinence, and treatment response to incontinence.
  7. Qmax and PVR
  8. PSA in the 2 months visit, then annually as per standard of care
  9. Serum creatinine level if indicated as standard of care
  10. Repeat cystoscopy and/or ultrasound if indicated as standard of care
* Researchers will collect patients' data and present initial results at 5 years and will continue collecting data after the initial reporting for future follow up studies.

Number of Patients to be enrolled:

Investigators will enroll at least 140 patients in the middle-lobe only PVP group and at least 140 patients in the complete PVP group.

Study Duration:

The study recruitment will continue until reaching the target sample size. Follow up the patients will continue until at least 5 years. Data will be collected beyond 5 years for possible future studies if the patient agrees up to 10 years.

Study Conduct:

Description of Activities:

* Research team will recruit patients from clinical encounters, including clinic, cystoscopy.
* If the patient meets the inclusion and exclusion criteria, the patient will be asked if he wants to participate in this study.
* If he agrees, the patient will sign the informed consent and fill the questionnaires.
* Patients will be allocated into either group based on intraoperative findings
* Post-operative care and follow up will be carried out based on the study protocol.

Patient Discontinuation from the Study:

If a patient wants to withdraw from the study after signing the consent form and before the procedure, the patient will not be included, and standard PVP procedure will be carried out as a standard of care.

If a patient after completing the procedure wishes to withdraw from the study, we will discontinue his follow up but we will keep the data up to his discontinuation. the withdrawals will be counted, and we will ask the patient about the reason for withdrawal if he wishes, which will be documented in the research results. The follow up for such patients will continue as the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Adult males (18-year-old and more)
* Suffering bothersome LUTS or urinary retention secondary to BPH
* Cystoscopic examination documenting the predominant middle lobe prostatic adenoma that is considered to be the primary cause of BOO.

Exclusion Criteria:

* Patients neurogenic lower urinary tract dysfunction (Neurogenic Bladder)
* Not competent to give consent and/or inability to provide answers to the questionnaire
* Patient who refuse to participate in the study
* Patients without a median lobe
* Patients who have a large prostate (more than 120 g on trans-abdominal ultrasound prostate sizing).
* Patients who have renal impairment secondary to BPH
* Patients with proven or suspicion of prostate cancer based on clinical examination and/or PSA level
* Patients with refractory hematuria secondary to BPH
* Patients with urethral strictures
* Patients with bladder cancer
* Patients with history of pelvic radiotherapy

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Inability to void | 3 months
  incidence of inability to void that needs surgical intervention after Middle lobe only PVP compared to complete PVP
IPSS | 3 months to 5 years
  The difference in international prostate symptoms score (IPSS) pre and post interventions and compare it between groups
Qmax | 3 months to 5 years
  The difference in Maximal flow rate (Qmax) pre and post interventions and compare it between groups
PVR | 3 months to 5
  The difference in Post void residual pre and post interventions and compare it between groups
MSHQ-EJD | 3 months to 5 years
  The difference in Male sexual health questionnaire ejaculatory dysfunction (MSHQ-EjD) pre and post interventions and compare it between groups

SECONDARY OUTCOMES:
Efficaciy of MLO based on prostate size, PSA, IPP and/or lateral lobes adenine | 3 months to 5 years
  Subset analysis of the efficacy and change of treatment urodynamic outcomes based prostate size, PSA, and presence or absence of IPP and/or lateral lobe adenomas.
additional treatment | 3 months to 5 years
  Documenting of the need for additional treatment of interventions
bleeding | 3 months
  The documentation of the blood loss and the need for blood transfusion
rate of patients with prominent middle lobe who needs MLO PVP | 3 months to 5 years
  • Determination of the rate of patients that initially thought to have middle lobe predominant obstruction on pre-operative cystoscopy but needed complete PVP due to inadequate removal of adenoma after completing middle-lobe only PVP
Erectile dysfunction MSHQ | 3 months to 5 years
  • Documentation of changes in erectile function using the Male sexual health questionnaire (MSHQ) Male Sexual Health Questionnaire (MSHQ)
additional medications | 3 months to 5 years
  • Determination the need to be on BPH medication in both groups at each follow up visit.
dysuria | 3 months to 5 years
  • Documentation of the presence of dysuria and compare it between the groups.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nickel JC, Aaron L, Barkin J, Elterman D, Nachabe M, Zorn KC. Canadian Urological Association guideline on male lower urinary tract symptoms/benign prostatic hyperplasia (MLUTS/BPH): 2018 update. Can Urol Assoc J. 2018 Oct;12(10):303-312. doi: 10.5489/cuaj.5616. No abstract available. PMID 30332601
- [Background] May F, Hartung R. Surgical atlas. Transurethral resection of the prostate. BJU Int. 2006 Oct;98(4):921-34. doi: 10.1111/j.1464-410X.2006.06474.x. No abstract available. PMID 16978302
- [Background] Zorn KC, Liberman D. GreenLight 180W XPS photovaporization of the prostate: how I do it. Can J Urol. 2011 Oct;18(5):5918-26. PMID 22018158
- [Background] Luo GC, Foo KT, Kuo T, Tan G. Diagnosis of prostate adenoma and the relationship between the site of prostate adenoma and bladder outlet obstruction. Singapore Med J. 2013 Sep;54(9):482-6. doi: 10.11622/smedj.2013168. PMID 24068054
- [Background] Gul Z, Chughtai B, Te AE, Thomas D, Kaplan SA. Ejaculatory Preserving Middle Lobe Onl-Transurethral Resection and Vaporization of the Prostate: 12-Year Experience. Urology. 2019 Dec;134:199-202. doi: 10.1016/j.urology.2019.07.042. Epub 2019 Sep 26. PMID 31563537
- [Background] Cornu JN, Ahyai S, Bachmann A, de la Rosette J, Gilling P, Gratzke C, McVary K, Novara G, Woo H, Madersbacher S. A Systematic Review and Meta-analysis of Functional Outcomes and Complications Following Transurethral Procedures for Lower Urinary Tract Symptoms Resulting from Benign Prostatic Obstruction: An Update. Eur Urol. 2015 Jun;67(6):1066-1096. doi: 10.1016/j.eururo.2014.06.017. Epub 2014 Jun 25. PMID 24972732
- [Background] Rassweiler J, Teber D, Kuntz R, Hofmann R. Complications of transurethral resection of the prostate (TURP)--incidence, management, and prevention. Eur Urol. 2006 Nov;50(5):969-79; discussion 980. doi: 10.1016/j.eururo.2005.12.042. Epub 2006 Jan 30. PMID 16469429